CLINICAL TRIAL: NCT05560906
Title: Study of Virus-specific Lymphocytic Cell Populations in Non-invasive Nasal Mucosa Samples of MIS-C Patients, and Intra-population Shifts in Inflammatory Tissues in the Acute Phase of MIS-C and in Health
Brief Title: Study of Virus-specific Lymphocytic Cell Populations in Non-invasive Nasal Mucosa Samples of MIS-C Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Collaborators: Erasmus Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Wojciech Feleszko, Associate Professor, MD., PhD, Medical University of Warsaw
Other Study IDs: NAWA015
Record Dates: First submitted 2022-09-13; First posted 2022-09-30 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: MIS-C Associated With COVID-19; COVID-19
Keywords: leukocytes; immunophenotype; nasal mucosa; curettage
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — Peripherial blood mononuclear cell samples Whole blood samples Leukocytes obtained during nasal mucosa curettage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Healthy patients under 18 years of age.
- MIS-C group: Patients with MIS-C diagnosed, based on WHO diagnostic criteria.

SUMMARY:
The aim of the study is to make an accurate assessment of immune cells obtained from nasal mucosa and peripherial blood of MIS-C patients during the disease and the period of health.

DETAILED DESCRIPTION:
The study will consist of two parts. Initially, it will be of a cross-cutting comparative nature, when a group of healthy patients (control group) and a group of patients diagnosed with MIS-C/PIMS syndrome are compared with each other, based on nasal curettage swabs and peripheral blood, before the inclusion of systemic anti-inflammatory treatment (study group). In addition, an observation of the research group will be carried out, during which swabs and peripheral blood will be taken at two more control points.

ELIGIBILITY:
Inclusion Criteria:

* MIS-C diagnosis based of WHO diagnostic criteria.

Exclusion Criteria:

* immunosuppressive treatment received up to 3 months before
* intranasal drugs received up to 7 days before
* COVID-19 vaccination
* no consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Acute MIS-C patients who have not received any treatment that could have altered nasal mucosa leukocyte composition. Samples will be collected from them at three time points.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in leukocyte subpopulations in nasal mucosa and peripherial blood during MIS-C and convalescence. | Three clinical timepoints: (i) baseline (preferably before immunomodulatory treatment), (ii) convalescence, after major symptoms resolution (1 week +/-2 days after treatment introduction), (iii) outpatient control visit (6 weeks after hospital discharge)
  The cellular subpopulations will be characterized and clustered using prepared immunomarker array.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Feleszko, MD., PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Pediatric teaching clinical hospital, Warsaw Medical University, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Clinical data of study patients could be shared upon other researchers' request.
Supporting Information: CSR
Time Frame: After study patient data is processed.
Access Criteria: Upon researcher's personal request.

REFERENCES:
- [Background] Radia T, Williams N, Agrawal P, Harman K, Weale J, Cook J, Gupta A. Multi-system inflammatory syndrome in children & adolescents (MIS-C): A systematic review of clinical features and presentation. Paediatr Respir Rev. 2021 Jun;38:51-57. doi: 10.1016/j.prrv.2020.08.001. Epub 2020 Aug 11. PMID 32891582
- [Background] Pawar R, Gavade V, Patil N, Mali V, Girwalkar A, Tarkasband V, Loya S, Chavan A, Nanivadekar N, Shinde R, Patil U, Lakshminrusimha S. Neonatal Multisystem Inflammatory Syndrome (MIS-N) Associated with Prenatal Maternal SARS-CoV-2: A Case Series. Children (Basel). 2021 Jul 2;8(7):572. doi: 10.3390/children8070572. PMID 34356552
- [Background] Whittaker E, Bamford A, Kenny J, Kaforou M, Jones CE, Shah P, Ramnarayan P, Fraisse A, Miller O, Davies P, Kucera F, Brierley J, McDougall M, Carter M, Tremoulet A, Shimizu C, Herberg J, Burns JC, Lyall H, Levin M; PIMS-TS Study Group and EUCLIDS and PERFORM Consortia. Clinical Characteristics of 58 Children With a Pediatric Inflammatory Multisystem Syndrome Temporally Associated With SARS-CoV-2. JAMA. 2020 Jul 21;324(3):259-269. doi: 10.1001/jama.2020.10369. PMID 32511692
- [Background] Verdoni L, Mazza A, Gervasoni A, Martelli L, Ruggeri M, Ciuffreda M, Bonanomi E, D'Antiga L. An outbreak of severe Kawasaki-like disease at the Italian epicentre of the SARS-CoV-2 epidemic: an observational cohort study. Lancet. 2020 Jun 6;395(10239):1771-1778. doi: 10.1016/S0140-6736(20)31103-X. Epub 2020 May 13. PMID 32410760
- [Background] Godfred-Cato S, Bryant B, Leung J, Oster ME, Conklin L, Abrams J, Roguski K, Wallace B, Prezzato E, Koumans EH, Lee EH, Geevarughese A, Lash MK, Reilly KH, Pulver WP, Thomas D, Feder KA, Hsu KK, Plipat N, Richardson G, Reid H, Lim S, Schmitz A, Pierce T, Hrapcak S, Datta D, Morris SB, Clarke K, Belay E; California MIS-C Response Team. COVID-19-Associated Multisystem Inflammatory Syndrome in Children - United States, March-July 2020. MMWR Morb Mortal Wkly Rep. 2020 Aug 14;69(32):1074-1080. doi: 10.15585/mmwr.mm6932e2. PMID 32790663
- [Background] Harwood R, Allin B, Jones CE, Whittaker E, Ramnarayan P, Ramanan AV, Kaleem M, Tulloh R, Peters MJ, Almond S, Davis PJ, Levin M, Tometzki A, Faust SN, Knight M, Kenny S; PIMS-TS National Consensus Management Study Group. A national consensus management pathway for paediatric inflammatory multisystem syndrome temporally associated with COVID-19 (PIMS-TS): results of a national Delphi process. Lancet Child Adolesc Health. 2021 Feb;5(2):133-141. doi: 10.1016/S2352-4642(20)30304-7. Epub 2020 Sep 18. PMID 32956615
- [Background] Gruber CN, Patel RS, Trachtman R, Lepow L, Amanat F, Krammer F, Wilson KM, Onel K, Geanon D, Tuballes K, Patel M, Mouskas K, O'Donnell T, Merritt E, Simons NW, Barcessat V, Del Valle DM, Udondem S, Kang G, Gangadharan S, Ofori-Amanfo G, Laserson U, Rahman A, Kim-Schulze S, Charney AW, Gnjatic S, Gelb BD, Merad M, Bogunovic D. Mapping Systemic Inflammation and Antibody Responses in Multisystem Inflammatory Syndrome in Children (MIS-C). Cell. 2020 Nov 12;183(4):982-995.e14. doi: 10.1016/j.cell.2020.09.034. Epub 2020 Sep 14. PMID 32991843
- [Background] Okarska-Napierala M, Mandziuk J, Feleszko W, Stelmaszczyk-Emmel A, Panczyk M, Demkow U, Kuchar E. Recurrent assessment of lymphocyte subsets in 32 patients with multisystem inflammatory syndrome in children (MIS-C). Pediatr Allergy Immunol. 2021 Nov;32(8):1857-1865. doi: 10.1111/pai.13611. Epub 2021 Aug 11. PMID 34331778
- [Background] Roukens AHE, Pothast CR, Konig M, Huisman W, Dalebout T, Tak T, Azimi S, Kruize Y, Hagedoorn RS, Zlei M, Staal FJT, de Bie FJ, van Dongen JJM, Arbous SM, Zhang JLH, Verheij M, Prins C, van der Does AM, Hiemstra PS, de Vries JJC, Janse JJ, Roestenberg M, Myeni SK, Kikkert M, Yazdanbakhsh M, Heemskerk MHM, Smits HH, Jochems SP; in collaboration with BEAT-COVID group; in collaboration with COVID-19 LUMC group. Prolonged activation of nasal immune cell populations and development of tissue-resident SARS-CoV-2-specific CD8+ T cell responses following COVID-19. Nat Immunol. 2022 Jan;23(1):23-32. doi: 10.1038/s41590-021-01095-w. Epub 2021 Dec 22. PMID 34937933